CLINICAL TRIAL: NCT04631133
Title: LISA Post Market Clinical Follow-Up Study:Post Marketing Prospective Documentation of Clinical Outcomes (Post-operative, Safety and Performance) After Lumbar Dynamic Stabilization Surgery With LISA Implant
Brief Title: LISA Post Market Clinical Follow-Up Study: Documentation of Clinical Outcomes After Surgery With LISA Implant
Acronym: LISA-PMCF
Status: Recruiting | Type: Observational
Sponsor: BACKBONE (Industry)
Responsible Party: Sponsor
Other Study IDs: DHF-111-PMCF1
Record Dates: First submitted 2020-11-02; First posted 2020-11-17 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Chronic Low-back Pain; Herniated Disc; Degenerative Disc Disease; Lumbar Canal Stenosis
Keywords: Chronic Low-back Pain; Herniated Disc; Degenerative Disc Disease; Lumbar Canal Stenosis; Dynamic Stabilization Implants; Post-Market Clinical Follow-Up Study
MeSH Terms: conditions — Intervertebral Disc Displacement; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with low-back pain and degenerative lesions of grade II, III, IV (Pfirrmann MRI class): Participants with low-back pain that accompanies degenerative lesions of grade II, III and IV (Pfirrmann MRI classification)
  Interventions: Device: Lumbar Implant for Stiffness Augmentation (LISA)

INTERVENTIONS:
Device: Lumbar Implant for Stiffness Augmentation (LISA) — The LISA Posterior Dynamic Stabilization System is intended to treat low-back pain that accompanies degenerative lesions of grade II, III and IV (Pfirrmann MRI classification).

SUMMARY:
The study is a post-market surveillance study of the Lumbar Implant for Stiffness Augmentation (LISA), a medical device, which is used to treat low-back pain that accompanies degenerative lesions of grades II, III, and IV (Pfirrmann MRI classification). "Post-market" means the device (i.e. the LISA implant) being used in this study has already obtained CE certification and is commercially available for use in the European market.

The LISA device consists of 3 components: A PEEK interspinous spacer, a polyester band, and a titanium blocker. The spacer is positioned between two adjacent spinous processes, the band is belted around the spinous processes and through the spacer, and the blocker is used to lock the band inside the spacer.

Medical Device manufacturers conduct "post-market" clinical studies in order to continuously evaluate the product scientifically and to comply with legal and ethical obligations. With these studies, the long-term safety as well as performance of their medical devices are assessed.

This study, which is initiated and sponsored by BACKBONE (LISA designer, developer, manufacturer and marketer), aims to evaluate the long-term safety and performance of the LISA implant for the treatment of lumbar degenerative disease and to evaluate the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients Patient ≥18 years of age
* Patients with low-back pain caused by degenerative lesions of grade II, III and IV (Pfirrmann MRI classification)
* Failed conservative treatment for low back pain conducted for at least 6 months

Exclusion Criteria:

* Stage V degenerative disk lesions in Pfirrmann's MRI classification
* Spondylolisthesis
* Osteoporosis
* Non-specific back pain
* Modic 2 and Modic 3 changes
* L5/S1 segments affected
* Local or general infections that may compromise the surgical goals
* Major local inflammatory phenomena
* Pregnant and lactating Women
* Immunosuppressive diseases
* Bone immaturity
* Severe mental illnesses
* Bone metabolism diseases that may compromise the mechanical support expected from this type of implant
* Patient with worker's compensation, under litigation or on disability benefits
* Excessive physical activities
* Patients deprived of their liberty in accordance with respective national regulations
* Protected patients or patients not in a position to declare his or her consent in accordance with respective national regulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must meet all inclusion criteria, and none of the exclusion criteria as described in the instructions for use of the LISA implant.
  The Lumbar Implant for Stiffness Augmentation, LISA, treats low-back pain that accompanies degenerative lesions of grade II, III and IV (Pfirrmann MRI classification).
Sampling Method: Non-Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2019-04-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
LISA implant survival rate 2 years after surgery defined as successful LISA implantation without reoperation, revision, or removal/ ODI change between pre-operative assessment and 2 years follow-up (FU)/ 1ary endpoint will also be evaluated at 1-year FU | 24-months post surgery; 12-months post surgery

SECONDARY OUTCOMES:
LISA implant survival rate defined as successful LISA implantation without reoperation, revision, or removal | 3-months post surgery; 6-months post surgery; 48-months post surgery; 72-months post surgery
Duration of the surgery | Perioperative
Duration of the implant placement | Perioperative
Amount of blood loss | Perioperative
Scoring of the surgical technique assessed by a 14-items question | Perioperative
  14 steps of the surgical technique are rated from 0 to 7; 0 being considered as very easy and 7 being considered as very difficult
Number of hospitalization days | 3-months post surgery
Time to return to normal activity (working) depending on the patient's profession (blue collar, white collar) | 3-months post surgery
Number of patients with reoperations/ revision or removal at the operative level or on adjacent levels relating to the device and not the pathology/ implant breakage (polyester band rupture) | 3-months post surgery; 6-months post surgery; 12-months post surgery; 24-months post surgery; 48-months post surgery; 72-months post surgery
Number of patients with migration or rupture of any implant component (Polyester band loose)/ major unanticipated device related complications/ post-operative scapular pain/ recurrence of the initial symptoms/ degeneration of the adjacent segments | 3-months post surgery; 6-months post surgery; 12-months post surgery; 24-months post surgery; 48-months post surgery; 72-months post surgery
Number of patients with superficial infection/ dural injury/ bone fracture or bone erosion anywhere implant is in contact with the anatomy/ Any other procedure or device related adverse events | 3-months post surgery; 6-months post surgery; 12-months post surgery; 24-months post surgery; 48-months post surgery; 72-months post surgery
Oswestry Disability Index (ODI) to assess limitations of various activities of daily living. | Pre-operative
Change from baseline in Oswestry Disability Index at 3 months | 3-months post surgery
  Oswestry Disability Index (ODI) is used to assess limitations of various activities of daily living.
Change from baseline in Oswestry Disability Index at 6 months | 6-months post surgery
  Oswestry Disability Index (ODI) is used to assess limitations of various activities of daily living.
Change from baseline in Oswestry Disability Index at 48 months | 48-months post surgery
  Oswestry Disability Index (ODI) is used to assess limitations of various activities of daily living.
Change from baseline in Oswestry Disability Index at 72 months | 72-months post surgery
  Oswestry Disability Index (ODI) is used to assess limitations of various activities of daily living.
Visual Analogue Scale (VAS) to assess back pain | Pre-operative
  Patients rate their back pain from 0 to 10, "0" meaning "No pain at all" and "10" meaning "the worst pain ever possible"
Change from baseline in Visual Analogue Scale (VAS) for back pain at 3 months | 3-months post surgery
Change from baseline in Visual Analogue Scale (VAS) for back pain at 6 months | 6-months post surgery
Change from baseline in Visual Analogue Scale (VAS) for back pain at 12 months | 12-months post surgery
Change from baseline in Visual Analogue Scale (VAS) for back pain at 24 months | 24-months post surgery
Change from baseline in Visual Analogue Scale (VAS) for back pain at 48 months | 48-months post surgery
Change from baseline in Visual Analogue Scale (VAS) for back pain at 72 months | 72-months post surgery
Visual Analogue Scale (VAS) to assess right leg pain | Pre-operative
  Patients rate their right leg pain from 0 to 10, "0" meaning "No pain at all" and "10" meaning "the worst pain ever possible"
Change from baseline in Visual Analogue Scale (VAS) for right leg pain at 3 months | 3-months post surgery
Change from baseline in Visual Analogue Scale (VAS) for right leg pain at 6 months | 6-months post surgery
Change from baseline in Visual Analogue Scale (VAS) for right leg pain at 12 months | 12-months post surgery
Change from baseline in Visual Analogue Scale (VAS) for right leg pain at 24 months | 24-months post surgery
Change from baseline in Visual Analogue Scale (VAS) for right leg pain at 48 months | 48-months post surgery
Change from baseline in Visual Analogue Scale (VAS) for right leg pain at 72 months | 72-months post surgery
Visual Analogue Scale (VAS) to assess left leg pain | Pre-operative
  Patients rate their left leg pain from 0 to 10, "0" meaning "No pain at all" and "10" meaning "the worst pain ever possible"
Change from baseline in Visual Analogue Scale (VAS) for left leg pain at 3 months | 3-months post-surgery
Change from baseline in Visual Analogue Scale (VAS) for left leg pain at 6 months | 6-months post-surgery
Change from baseline in Visual Analogue Scale (VAS) for left leg pain at 12 months | 12-months post-surgery
Change from baseline in Visual Analogue Scale (VAS) for left leg pain at 24 months | 24-months post-surgery
Change from baseline in Visual Analogue Scale (VAS) for left leg pain at 48 months | 48-months post-surgery
Change from baseline in Visual Analogue Scale (VAS) for left leg pain at 72 months | 72-months post-surgery
Patient satisfaction with treatment assessed by a 4-items question | 3-months post surgery; 6-months post surgery; 12-months post surgery; 24-months post surgery; 48-months post surgery; 72-months post surgery
  Patients rate their satisfaction with treatment choosing one of the following options: Very satisfied/Somewhat satisfied/Somewhat dissatisfied/Very Dissatisfied
Patient's recommendation for treatment assessed by a 4-items question | 3-months post surgery; 6-months post surgery; 12-months post surgery; 24-months post surgery; 48-months post surgery; 72-months post surgery
  Patient rate wether they would recommend the same treatment to a friend with the same condition, choosing one of the following options: Definitely YES/Probably YES/ Probably NO/ Definitely NOT
Patient's opinion related to the treatment assessed by a 6-items question | 3-months post surgery; 6-months post surgery; 12-months post surgery; 24-months post surgery; 48-months post surgery; 72-months post surgery
  Patient rate how effective was the treatment in eliminating the symptoms choosing one of the following options: "very effective, relieved all the symptoms", "moderately effective", "somewhat effective", "somewhat ineffective", "moderately ineffective", "very ineffective, did not relieve or lessen the symptoms"
Surgeon surgery outcome assessed by a 4-items question | 3-months post surgery; 6-months post surgery; 12-months post surgery; 24-months post surgery; 48-months post surgery; 72-months post surgery
  Surgeons rate the result of the surgery, choosing one of the following options: Excellent; Good; Fair; Poor
Segmental joints condition assessed thanks to radiological results (if available) | Pre-operative
Change from baseline in segmental joints condition at 3-months | 3-months post surgery
  Segmental joints condition are assessed thanks to radiological results (if available)
Change from baseline in segmental joints condition at 6-months | 6-months post surgery
  Segmental joints condition are assessed thanks to radiological results (if available)
Change from baseline in segmental joints condition at 12-months | 12-months post surgery
  Segmental joints condition are assessed thanks to radiological results (if available)
Change from baseline in segmental joints condition at 24-months | 24-months post surgery
  Segmental joints condition are assessed thanks to radiological results (if available)
Change from baseline in segmental joints condition at 48-months | 48-months post surgery
  Segmental joints condition are assessed thanks to radiological results (if available)
Change from baseline in segmental joints condition at 72-months | 72-months post surgery
  Segmental joints condition are assessed thanks to radiological results (if available)
Narrowness of the spinal canal assessed thanks to radiological results (if available) | Pre-operative
Change from baseline in narrowness of the spinal canal at 3 months | 3-months post surgery
  Narrowness of the spinal canal is assessed thanks to radiological results (if available)
Change from baseline in narrowness of the spinal canal at 6 months | 6-months post surgery
  Narrowness of the spinal canal is assessed thanks to radiological results (if available)
Change from baseline in narrowness of the spinal canal at 12 months | 12-months post surgery
  Narrowness of the spinal canal is assessed thanks to radiological results (if available)
Change from baseline in narrowness of the spinal canal at 24 months | 24-months post surgery
  Narrowness of the spinal canal is assessed thanks to radiological results (if available)
Change from baseline in narrowness of the spinal canal at 48 months | 48-months post surgery
  Narrowness of the spinal canal is assessed thanks to radiological results (if available)
Change from baseline in narrowness of the spinal canal at 72 months | 72-months post surgery
  Narrowness of the spinal canal is assessed thanks to radiological results (if available)
Foraminal compression assessed thanks to radiological results (if available) | Pre-operative
Change from baseline in foraminal compression at 3 months | 3-months post-surgery
  Foraminal compression is assessed thanks to radiological results (if available)
Change from baseline in foraminal compression at 6 months | 6-months post-surgery
  Foraminal compression is assessed thanks to radiological results (if available)
Change from baseline in foraminal compression at 12 months | 12-months post-surgery
  Foraminal compression is assessed thanks to radiological results (if available)
Change from baseline in foraminal compression at 24 months | 24-months post-surgery
  Foraminal compression is assessed thanks to radiological results (if available)
Change from baseline in foraminal compression at 48 months | 48-months post-surgery
  Foraminal compression is assessed thanks to radiological results (if available)
Change from baseline in foraminal compression at 72 months | 72-months post-surgery
  Foraminal compression is assessed thanks to radiological results (if available)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Pointillart, Principal Investigator — Pellegrin University Hospital Center
Locations (5):
- Elective Surgery Center, Silkeborg Regional Hospital, Silkeborg, Denmark
- France (3):
  - Pellegrin University Hospital Center, Bordeaux
  - Saint-Charles Clinic, Lyon
  - Pitié-Salpêtrière University Hospital Center, Paris
- Asklepios Stadtklinik, Bad Wildungen, Bad Wildungen, Germany